CLINICAL TRIAL: NCT02083419
Title: Study of the Effects of Cardiac Resynchronization Therapy (CRT) and Left Ventricular Assist Devices (LVAD) Therapy
Brief Title: Cardiac Resynchronization Therapy (CRT) and Left Ventricular Assist Devices (LVAD) Therapy
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201300694
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Heart Failure
Keywords: Left Ventricular Assist Devices (LVAD); Cardiac Resynchronization Devices (CRT)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LVAD CRT: The following procedures will be performed: limited echocardiogram, an adjustment to the CRT device's programmed settings, follow-up in 30 days to adjust the CRT device's programmed settings. In addition, quality of life questionnaires will be filled out and a 6 minute walk test will be completed.
  Interventions: Device: LVAD CRT

INTERVENTIONS:
Device: LVAD CRT — The following procedures will be performed: limited echocardiogram, an adjustment to the CRT device's programmed settings, follow-up in 30 days to adjust the CRT device's programmed settings. In addition, quality of life questionnaires will be filled out and a 6 minute walk test will be completed.

SUMMARY:
Cardiac resynchronization therapy (CRT) or biventricular pacing is a useful treatment for heart failure and those suffering from arrhythmias. The purpose of this research study is to determine the effect left-ventricular pacing has on patients who have a ventricular assist device.

DETAILED DESCRIPTION:
As part of the study participation the following two visits will be completed as listed below.

Baseline Visit: The following procedures will be conducted at this visit:

* Review of past medical history and medical records;
* A limited echocardiogram will be performed. This is a test that uses ultrasound to evaluate the size of the heart and how well the heart is pumping blood.
* The investigators will use a computer-like device, called a programmer, that "talks" to the CRT device using radio signals or by using wanded telemetry to adjust the CRT device's programmed settings. The left ventricular lead of your device will be turned off. The defibrillator will continue to function and back-up pacing will continue if needed.
* Complete the Kansas City Cardiomyopathy Questionnaire (KCCQ).
* A 6 minute walk test will be done.

Regularly Scheduled Clinic Visit: At the next regularly scheduled Left Ventricular Assist Devices (LVAD) clinic visit, approximately 4 weeks after the baseline visit, the following procedures will be done:

* A second limited echocardiogram.
* The investigator will use a computer-like device, called a programmer, that "talks" to the CRT device using radio signals or by using a wand to obtain a report that will give the current program settings and any heart rhythm events that have occurred since the last CRT device was checked. Once the information from the CRT is obtained, the study doctor will reprogram the device to its original settings.
* Complete the Kansas City Cardiomyopathy Questionnaire (KCCQ).
* A 6 minute walk test will be done.

ELIGIBILITY:
Inclusion Criteria:

* Presence of LVAD support and CRT device with working LV lead in patients > 18years of age
* Left ventricular pacing at time of enrollment

Exclusion Criteria:

* LV lead dysfunction
* Prior AV node ablation
* Presence of total heart block
* Presence of significant bradycardia/lack of underlying rhythm
* Inability to complete 6 minute walk test
* Inability to return to clinic for repeat assessment
* Any LVAD programmed speed change within the prior 30 days
* Any CRT programming changes within the prior 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with ventricular dysfunction, dyssynchrony, functional capacity presence of arrhythmia. LVAD patients undergo 6 minute walk testing and complete a quality of life questionnaire routinely as part of their care on our LVAD clinic. Additionally, periodic echcoardiography is obtained to determine LVAD dynamics and ventrocular dimensions. We will utilize this information for our study, as well as information from their cardiac resynchronization devices, which is part of routine care for patietns with pacemakers and defibrillators.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Change in echocardiographic parameters | Change in baseline to 30 days
  A comparison of the echocardiogram completed at enrollment and at 30 days.
6 minute walk distance | Change in baseline to 30 days
  A trained staff member will supervise participants in the completion of a 6 minute walk test. They will be instructed to walk on a level surface, on a clearly marked indoor course. heart rate and oxygen level will be monitored. The total distance completed at the end of 6 minutes will be noted.
Quality of Life | Change in baseline to 30 days
  A comparison of the questionnaires completed at enrollment and at 30 days.
Number of Ventricular Tachycardia Episodes | Change in baseline to 30 days
  At baseline and again at 30 days CRT device interrogation will be done to count the number of ventricular tachycardia episodes with LV pacing on and off.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Ahmed, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States